CLINICAL TRIAL: NCT02446821
Title: Evaluation of the Effectiveness, Safety and Tolerability of the ContraMed VeraCept Intrauterine Copper Contraceptive for Long-Acting Reversible Contraception
Brief Title: Evaluation of ContraMed VeraCept Intrauterine Copper Contraceptive for Long Acting Reversible Contraception
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sebela Women's Health Inc. (Industry)
Collaborators: Premier Research (Other)
Responsible Party: Sponsor
Organization: Sebela Pharmaceuticals Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMDOC-0008
Record Dates: First submitted 2015-04-24; First posted 2015-05-18 (Estimated); Results first posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Contraception

STUDY DESIGN:
Intervention Model Description: VeraCept intrauterine contraceptive device
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- VeraCept IUD System (Experimental): All women will receive VeraCept.
  Interventions: Drug: VeraCept

INTERVENTIONS:
Drug: VeraCept — IUD placement of VeraCept

SUMMARY:
Prospective, multi-center, single-arm, open-label, Phase II clinical study to evaluate the effectiveness, device placement, safety, and tolerability of VeraCept to support commencing a Phase III Clinical Study

DETAILED DESCRIPTION:
Up to 250 subjects will be consented, screened and have VeraCept placed, with a goal to have 2240 evaluable cycles at 12 months. It is planned that 225 of the 250 subjects will be within the 18-35 year age range, with a total of 2015 evaluable cycles. The remaining 25 subjects will be within the 35-40 year age range.

Follow-up: Physical assessment (office visit) will occur at weeks 6, 13, 26 and 52 after placement, with monthly telephone contact. For those subjects who wish to continue study device use after 12 months, follow-up office visits will occur every 6 months. Additional visits will be conducted if necessary for safety issues.

Follow-up after early study device removal:

Subjects requesting VeraCept removal to become pregnant will be followed to pregnancy or until the subject changes their mind about trying to get pregnant. All subjects in whom VeraCept is removed prior to 12 months, for any reason, will be required to use an alternative contraceptive for the first two weeks following removal. Progestin-only pills will be provided by the sponsor as a contraceptive option during this time unless the subject has a category 4 condition precluding their use.

Study Population: Pre-menopausal women ages 18 - 40, at risk for pregnancy, who are interested in using an intrauterine contraceptive for birth control will be eligible for this study. Subjects must provide written informed consent and meet the study subject selection criteria without any exclusions as outlined in the Clinical Investigation Plan (CIP).

Primary Effectiveness Outcome: The primary outcome measure is effectiveness, evaluated as the absence of pregnancy by 12 months, failure will be calculated by the Pearl Index.

Safety and Other Outcome

Measures: Safety and other outcome measures include:

Study Device Placement:

* Ease of placement
* Placement success

Safety:

* Serious Adverse Events
* Adverse Events

Tolerability:

* Bleeding and spotting patterns
* Discontinuation rate and reasons for discontinuation

ELIGIBILITY:
Inclusion Criteria:

1. Between 18-40 years of age at the time of study initiation;

   1.1 Enrollment will be targeted for 225 subjects aged 18-35 (for safety and effectiveness analyses) and an additional 25 subjects aged 36-40 (for safety only) (note: all subjects will be included in the analysis for device placement and tolerability);
2. Pre-menopausal, as determined by regular menstrual cycle (28 ± 5 days) for the last 3 months;

   2.1 Based on patient history, when not on hormonal contraceptives;
3. Sexually active with a male partner who has not had a vasectomy;
4. Reasonably expect to have to coitus at least once monthly during the study period.
5. Married or in a steady relationship (e.g., 3-6 months);
6. Seeking to avoid pregnancy for the next 12 months;
7. Willing to use the study device as the sole form of contraception;
8. Willing to accept a risk of pregnancy;
9. Normal PAP or ASC-US with negative high risk HPV test result within the appropriate screen timeframe, unless considered at risk;
10. Able and willing to comply with all study tests, procedures, assessment tools and follow-up; and
11. Able and willing to provide and document informed consent and Authorization for Release of Protected Health Information (PHI).

Exclusion Criteria:

1. Known or suspected pregnancy; or at risk for pregnancy from unprotected intercourse earlier in current cycle
2. Subject who anticipates separation from her partner for more than 1 cycle within the next 12 months;
3. A previously inserted IUD that has not been removed by the time VeraCept is placed;
4. History of previous IUD complications, such as perforation, expulsion, infection (pelvic inflammatory disease) or pregnancy with IUD in place;
5. Injection of hormonal contraceptive (e.g., Depo-Provera) within the last 10 months;

   5.1 Must have had 2 normal menstrual cycles since the last injection;
6. Planned use of any non-contraceptive estrogen, progesterone or testosterone any time during the 12 months of study participation;
7. Postpartum, prior to a minimum of 6 weeks or complete uterine involution;
8. Exclusively breastfeeding before return of menses; Lactating women will be excluded unless they have had two normal menstrual periods.

   8.1 Must have had 2 normal spontaneous menstrual cycles since delivery
9. Unexplained abnormal uterine bleeding (suspicious for serious condition), before evaluation; Immediately post-septic abortion or puerperal sepsis;
10. Severely heavy or painful menstrual bleeding;
11. Suspected or known cervical, uterine or ovarian cancer, or unresolved clinically significant abnormal pap smear requiring evaluation or treatment
12. Any history of gestational trophoblastic disease with or without detectable elevated ß-hCG levels, or related malignant disease;
13. Known anatomical abnormalities of the uterine cavity that may complicate IUD placement, such as:

    13.1 Submucosal uterine leiomyoma

    13.2 Asherman's syndrome

    13.3 Pedunculated polyps

    13.4 Bicornuate uterus

    13.5 Didelphus or uterine septa
14. Known anatomical abnormalities of the cervix such as severe cervical stenosis, prior trachelectomy or extensive conization that, in the opinion of the investigator would prevent cervical dilation and study device placement;
15. Current or recent (within the last 3 months) pelvic infection (cervix, endometrium, or fallopian tubes), or mucopurulent cervicitis;
16. High risk for STDs (e.g., multiple sexual partners);
17. Known or suspected AIDS;
18. Known intolerance or allergy to nickel or copper, including Wilson's Disease;
19. Currently participating or planning future participation in a research study of an investigational drug or device during the course of this investigational study;
20. Subject had VeraCept placed previously or had 2 attempts at placement;
21. Known or suspected alcohol or drug abuse within 12 months prior to the screening visit;
22. Any general health or behavioral condition that, in the opinion of the Investigator, could represent an increased risk for the subject or would render the subject less likely to provide the needed study information.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 286 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2019-03-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anita L Nelson, MD, Principal Investigator — University of California, Los Angeles
Locations (12):
- United States (12):
  - Essential Access Health (formerly California Family Health Council), Burbank, California
  - Essential Access Health (formerly California Family Health Council), Los Angeles, California
  - University of California Davis Health System, Sacramento, California
  - University of Colorado, Aurora, Colorado
  - Healthcare Clinical Data, Inc, Miami, Florida
  - Columbia University Medical Center, New York, New York
  - University of Cincinnati, Cincinnati, Ohio
  - Oregon Health and Sciences University, Portland, Oregon
  - Clinical Research of Philadelphia, Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Advanced Research Associates, Corpus Christi, Texas
  - University of Utah, Salt Lake City, Utah

REFERENCES:
- [Derived] Turok DK, Nelson AL, Dart C, Schreiber CA, Peters K, Schreifels MJ, Katz B; VeraCept Phase 2 Clinical Investigator Group. Efficacy, Safety, and Tolerability of a New Low-Dose Copper and Nitinol Intrauterine Device: Phase 2 Data to 36 Months. Obstet Gynecol. 2020 Apr;135(4):840-847. doi: 10.1097/AOG.0000000000003756. PMID 32168217

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | VeraCept IUD System
Started | 286
Completed | 218
Not Completed | 68
Not completed — Adverse Event | 28
Not completed — Withdrawal by Subject | 6
Not completed — Lost to Follow-up | 22
Not completed — other | 9
Not completed — insertion failure | 3

BASELINE CHARACTERISTICS:
Arm/Group | VeraCept IUD System
Number analyzed (Participants) | 286
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.1 (5.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 286
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 48
  Not Hispanic or Latino | 238
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3
  Asian | 19
  Native Hawaiian or Other Pacific Islander | 2
  Black or African American | 69
  White | 182
  More than one race | 0
  Unknown or Not Reported | 11

OUTCOME MEASURES:

1. Primary Outcome: The Primary Outcome Measure is Effectiveness as Calculated by the Pearl Index
Description: The Pearl Index is calculated as the number of on-treatment pregnancies per 100 woman-years of exposure. On-treatment pregnancy is defined as the estimated conception date being on or after the insertion date (must be a successful insertion) and no more than 7 days after the study drug is removed or expelled. One women year is defined as comprising thirteen 28-day cycles. A lower Pearl Index indicates greater contraceptive effectiveness.
Time Frame: 12 months
Population: Evaluation for Pregnancy Population
Measure: Number (95% Confidence Interval); unit: Pearl Index
Arm/Group | VeraCept IUD System
Number analyzed (Participants) | 248
Pearl Index
  All evaluable for pregnancy subjects | 0.53 [0.01 to 2.93]
  evaluable for pregnancy subjects with at least one live birth: number analyzed (Participants) | 92
  evaluable for pregnancy subjects with at least one live birth | 1.41 [0.04 to 7.88]
  evaluable for pregnancy subjects never had live birth: number analyzed (Participants) | 156
  evaluable for pregnancy subjects never had live birth | 0.00 [0 to 3.08]

2. Secondary Outcome: VeraCept Placement Success
Description: The number and percentage of subjects with either a successful or unsuccessful placement will be summarized
Time Frame: Visit 1 (Day 1)/ VeraCept Placement
Population: Intent to Treat Population
Measure: Count of Participants; unit: Participants
Arm/Group | VeraCept IUD System
Number analyzed (Participants) | 286
Participants
  successfully placed on first attempt | 267
  successfully placed on second attempt | 18
  not successfully placed | 3

3. Secondary Outcome: Ease of VeraCept Placement
Description: Ease of placement of the VeraCept was assessed by the clinician immediately following device placement. The clinician rated the ease of placement using the following options: "Very Easy," "Easy," "Neither Easy nor Hard," "Hard," or "Very Hard." This rating was based on the clinician's experience during the placement procedure.
Time Frame: Visit 1 (Day 1)/ VeraCept Placement
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | VeraCept IUD System
Number analyzed (Participants) | 283
Participants
  Very Easy | 173
  Easy | 86
  Neither Easy nor Hard | 11
  Hard | 8
  Very Hard | 5

4. Secondary Outcome: Bleeding and Spotting Patterns (Number of Bleeding and/or Spotting Days Per Cycle)
Description: Bleeding and spotting patterns will be summarized for the first year of treatment (Cycle 1 to Cycle 13) by the mean number of days in each 28-day cycle with bleeding or spotting, bleeding only, and spotting only
Time Frame: Cycle 1 to Cycle 13 (post IUD placement). Each cycle is 28 days.
Population: The Evaluable for Cycle Control (ECYC) Population includes subjects who provided bleeding-related diary data. The number of participants reported for each cycle reflects the number of ECYC subjects who submitted bleeding-related diary data during that specific cycle.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | VeraCept IUD System
Number analyzed (Participants) | 275
Days
  Cycle 1 : bleeding or spotting: number analyzed (Participants) | 274
  Cycle 1 : bleeding or spotting | 11.2 (5.83)
  Cycle 1 : bleeding only: number analyzed (Participants) | 274
  Cycle 1 : bleeding only | 7.6 (4.35)
  Cycle 1 : spotting only: number analyzed (Participants) | 274
  Cycle 1 : spotting only | 3.6 (3.71)
  Cycle 2 : bleeding or spotting: number analyzed (Participants) | 264
  Cycle 2 : bleeding or spotting | 8.1 (4.22)
  Cycle 2 : bleeding only: number analyzed (Participants) | 264
  Cycle 2 : bleeding only | 5.8 (3.29)
  Cycle 2 : spotting only: number analyzed (Participants) | 264
  Cycle 2 : spotting only | 2.2 (2.61)
  Cycle 3 : bleeding or spotting: number analyzed (Participants) | 259
  Cycle 3 : bleeding or spotting | 7.8 (4.12)
  Cycle 3 : bleeding only: number analyzed (Participants) | 259
  Cycle 3 : bleeding only | 5.8 (3.02)
  Cycle 3 : spotting only: number analyzed (Participants) | 259
  Cycle 3 : spotting only | 2.0 (2.32)
  Cycle 4 : bleeding or spotting: number analyzed (Participants) | 251
  Cycle 4 : bleeding or spotting | 7.2 (3.62)
  Cycle 4 : bleeding only: number analyzed (Participants) | 251
  Cycle 4 : bleeding only | 5.3 (2.60)
  Cycle 4 : spotting only: number analyzed (Participants) | 251
  Cycle 4 : spotting only | 1.9 (2.38)
  Cycle 5 : bleeding or spotting: number analyzed (Participants) | 242
  Cycle 5 : bleeding or spotting | 7.0 (3.67)
  Cycle 5 : bleeding only: number analyzed (Participants) | 242
  Cycle 5 : bleeding only | 5.3 (2.70)
  Cycle 5 : spotting only: number analyzed (Participants) | 242
  Cycle 5 : spotting only | 1.8 (2.61)
  Cycle 6 : bleeding or spotting: number analyzed (Participants) | 244
  Cycle 6 : bleeding or spotting | 7.6 (4.60)
  Cycle 6 : bleeding only: number analyzed (Participants) | 244
  Cycle 6 : bleeding only | 5.6 (3.60)
  Cycle 6 : spotting only: number analyzed (Participants) | 244
  Cycle 6 : spotting only | 2.0 (2.76)
  Cycle 7 : bleeding or spotting: number analyzed (Participants) | 237
  Cycle 7 : bleeding or spotting | 7.1 (3.81)
  Cycle 7 : bleeding only: number analyzed (Participants) | 237
  Cycle 7 : bleeding only | 5.3 (2.89)
  Cycle 7 : spotting only: number analyzed (Participants) | 237
  Cycle 7 : spotting only | 1.8 (2.25)
  Cycle 8 : bleeding or spotting: number analyzed (Participants) | 227
  Cycle 8 : bleeding or spotting | 6.9 (3.83)
  Cycle 8 : bleeding only: number analyzed (Participants) | 227
  Cycle 8 : bleeding only | 5.3 (2.94)
  Cycle 8 : spotting only: number analyzed (Participants) | 227
  Cycle 8 : spotting only | 1.6 (2.03)
  Cycle 9 : bleeding or spotting: number analyzed (Participants) | 223
  Cycle 9 : bleeding or spotting | 7.1 (4.00)
  Cycle 9 : bleeding only: number analyzed (Participants) | 223
  Cycle 9 : bleeding only | 5.3 (2.84)
  Cycle 9 : spotting only: number analyzed (Participants) | 223
  Cycle 9 : spotting only | 1.7 (2.39)
  Cycle 10 : bleeding or spotting: number analyzed (Participants) | 221
  Cycle 10 : bleeding or spotting | 7.0 (3.75)
  Cycle 10 : bleeding only: number analyzed (Participants) | 221
  Cycle 10 : bleeding only | 5.2 (2.90)
  Cycle 10 : spotting only: number analyzed (Participants) | 221
  Cycle 10 : spotting only | 1.7 (2.37)
  Cycle 11 : bleeding or spotting: number analyzed (Participants) | 219
  Cycle 11 : bleeding or spotting | 7.0 (3.57)
  Cycle 11 : bleeding only: number analyzed (Participants) | 219
  Cycle 11 : bleeding only | 5.3 (2.35)
  Cycle 11 : spotting only: number analyzed (Participants) | 219
  Cycle 11 : spotting only | 1.7 (2.40)
  Cycle 12 : bleeding or spotting: number analyzed (Participants) | 217
  Cycle 12 : bleeding or spotting | 7.0 (4.25)
  Cycle 12 : bleeding only: number analyzed (Participants) | 217
  Cycle 12 : bleeding only | 5.4 (3.25)
  Cycle 12 : spotting only: number analyzed (Participants) | 217
  Cycle 12 : spotting only | 1.7 (2.35)
  Cycle 13 : bleeding or spotting: number analyzed (Participants) | 211
  Cycle 13 : bleeding or spotting | 7.1 (4.75)
  Cycle 13 : bleeding only: number analyzed (Participants) | 211
  Cycle 13 : bleeding only | 5.2 (3.56)
  Cycle 13 : spotting only: number analyzed (Participants) | 211
  Cycle 13 : spotting only | 1.9 (2.96)

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | VeraCept IUD System
All-Cause Mortality (participants affected / at risk) | 0/286
Serious Adverse Events (participants affected / at risk) | 4/286
Other Adverse Events (participants affected / at risk) | 243/283
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VeraCept IUD System (N=286)
chronic tonsillitis (Infections and infestations) | 1 (1)
cellulitis (Infections and infestations) | 1 (1)
hyperbilirubinaemia (Blood and lymphatic system disorders) | 1 (1)
urinary tract infection (Infections and infestations) | 1 (1)
pelvic inflammatory disease (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VeraCept IUD System (N=283)
abdominal pain (Gastrointestinal disorders) | 38 (66)
abdominal pain lower (Gastrointestinal disorders) | 21 (43)
nausea (Gastrointestinal disorders) | 15 (15)
bacterial vaginosis (Infections and infestations) | 33 (43)
nasopharyngitis (Infections and infestations) | 61 (84)
upper respirtory tract infection (Infections and infestations) | 36 (51)
urinary tract infection (Infections and infestations) | 31 (35)
vulvovaginal mycotic infection (Infections and infestations) | 26 (31)
post procedural haemorrhage (Injury, poisoning and procedural complications) | 21 (21)
procedural pain (Injury, poisoning and procedural complications) | 99 (130)
back pain (Musculoskeletal and connective tissue disorders) | 30 (52)
headache (Nervous system disorders) | 39 (97)
dysmenorrhoea (Reproductive system and breast disorders) | 120 (234)
dyspareunia (Reproductive system and breast disorders) | 22 (24)
menorrhagia (Reproductive system and breast disorders) | 74 (177)
metrorrhagia (Reproductive system and breast disorders) | 35 (49)
pelvic pain (Reproductive system and breast disorders) | 35 (64)
uterine spasm (Reproductive system and breast disorders) | 24 (25)
vaginal discharge (Reproductive system and breast disorders) | 18 (20)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-09-19): https://cdn.clinicaltrials.gov/large-docs/21/NCT02446821/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-17): https://cdn.clinicaltrials.gov/large-docs/21/NCT02446821/SAP_001.pdf